CLINICAL TRIAL: NCT05592080
Title: Exploring Liver and Muscle Fat Content in Overweight and Obese Polycystic Ovary Syndrome Using Magnetic Resonance Imaging Technique
Brief Title: Exploring Liver and Muscle Fat Content Using MRI
Status: Completed | Type: Observational
Sponsor: Bing He (Other)
Responsible Party: Sponsor-Investigator, Bing He, Dr., Shengjing Hospital
Organization: Shengjing Hospital (Other)
Other Study IDs: 2022PS1008K
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pcos
  Interventions: Radiation: MRI
- non-pcos
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — MRI-mDIXON-Quant examinations, anthropometric measures, body composition, hormonal and biochemical assays were performed in all participants, and the liver fat fraction (LFF) and muscle fat fraction (MFF) represented the fat content in the liver and skeletal muscle, respectively.

SUMMARY:
The aim of our study was to compare the difference of fatty infiltration in liver and muscle using magnetic resonance imaging (MRI) between overweight as well as obese polycystic ovary syndrome (PCOS) cases and body mass index (BMI)-matched women without PCOS, identifying the possible influence factors.

ELIGIBILITY:
Inclusion Criteria:

(1) subjects with a body mass index (BMI) ≥ 24 kg/m2; (2) subjects aged between 18 and 40 years; (3) subjects who had not received any prescription or non-prescription drugs that affect insulin sensitivity or ovarian function, including hormonal contraceptives and metformin, within three months before the trial; (4) PCOS diagnosis fulfills the Rotterdam 2003 criteria phenotype B with hyperandrogenism (HA) and oligo-/anovulation [29]; (5) subjects who had not received medication that impacts lipid metabolism (fibrates, statins, antioxidants and diuretic) in the recent 3 months; (6) subjects who did not intend to become pregnant and use barrier contraception; (7) subjects who did not change their lifestyle, including physical activity and eating habits, during the study period.

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: (1) subjects with other causes of irregular menstrual cycles or androgen excess including hyperprolactinemia, uncontrolled thyroid disease, congenital adrenal hyperplasia, Cushing's disease, androgen secreting tumor, or pregnancy; (2)subjects with abnormal liver function test results (ALT level 2.5 times higher than the upper limit of the normal range); (3) subjects with renal insufficiency (eGFR < 60 ml/min/1.73 m2); (4) subjects with a history of chronic liver diseases such as alcoholic liver disease, viral hepatitis, autoimmune liver disease, drug-induced liver disease, genetic metabolic liver disease; (5) subjects experiencing alcoholism (weekly alcohol intake > 100 g) subjects experiencing smoking within the past 3 months and engaging in high-intensity exercise; (6) subjects with a history of cancer; (7) subjects with active infection; subjects who were pregnant or breastfeeding.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
liver fat fraction | 1 year
  liver fat fraction (LFF) represented the fat content in liver.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided